CLINICAL TRIAL: NCT05888220
Title: The Effect Of Warm Salt Water and Warm Water Bath Applied to Hands and Feet of Patients With Rheumatoid Arthritis on Pain, Fatigue, Sleep Quality and Functional Capacity,
Brief Title: Application of Warm Water and Warm Salt Water to Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, OKŞAN AKTAŞ, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/56
Record Dates: First submitted 2023-04-28; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis - Rheumatism
Keywords: pain,fatigue,sleep,functional status,rheumatoid arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- warm salt water group (Experimental): The patients were told how to prepare and apply the temperature and salt ratio of the water to be used in the hand and foot bath (280 grams of rock salt to 8 liters of water) with a demonstration method with video training. video tutorial tablet It was done in a quiet environment in the hospital, in a room with the patient and the researcher. The temperature of the water and the duration of application were determined based on research that previously examined the effectiveness of warm water and warm salt water baths in various patient groups. Bath hours were determined to be between 21:00 and 22:00 in order to prevent the patients from doing any activity after this application and to provide relaxation and rest after the bath. Starting 1 day after the training, each patient is at home for six weeks from 21:00 to He applied a warm salt water bath at 41°C for 20 minutes to his hands and feet three times a week between 21:00-22:00.
  Interventions: Other: warm salt water bath
- warm water group (Experimental): The patients were told how to prepare and apply the temperature of the water to be used in the hand and foot bath with video training and demonstration method. The video training was carried out using a tablet in a quiet environment in the hospital in a room with the patient and the researcher. The temperature of the water and the duration of application were determined based on research that previously examined the effectiveness of warm water and warm salt water baths in various patient groups. Bath hours were determined to be between 21:00 and 22:00 in order to prevent the patients from doing any activity after this application and to provide relaxation and rest after the bath. Starting 1 day after the training, each patient applied a 20-minute warm water bath at 41°C every other day, three times a week between 21:00 and 22:00 at home for six weeks, on their hands and feet.
  Interventions: Other: warm salt water bath
- control group (No Intervention): No intervention was made for the patients. Visual Analog Scale, Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, Pittsburgh Sleep Quality Index, Health Assessment Questionnaires were re-administered at the end of the sixth week in this group.

INTERVENTIONS:
Other: warm salt water bath — Warm water and warm salt water bath were applied to the hands and feet of the patients. It is a non-pharmacological intervention
  Other Names: warm water bath
  Arms: warm salt water group; warm water group

SUMMARY:
This pretest-posttest randomized controlled study aimed to determine the effect of warm salt water and warm water bath applied to the hands and feet on pain, fatigue, sleep quality, and functional capacity in patients with rheumatoid arthritis.

The study consisted of three groups. These groups consisted of two intervention groups and one control group. As a result of the power analysis, it was determined that 54 people should be reached. Visual Analog Scale, Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, Pittsburgh Sleep Quality Index, and Health Assessment Questionnaire were used in the study. Patients in intervention groups applied a 41°C warm salt and warm water bath three times a week for six weeks in line with the training given. The patients in the control group did not undergo any intervention other than routine treatment and care.

DETAILED DESCRIPTION:
The study was conducted at Gulhane Training and Research Hospital Rheumatology Polyclinic, in Turkey. The sample of the study consisted of 54 patients. Eighteen patients in the warm saltwater group were trained using the video demonstration method to make the intervention. Eighteen patients in the lukewarm water group were trained using the video demonstration method to make the intervention. Eighteen patients in the control group were not given any training other than their routine treatment and care. Each patient's pain, fatigue, sleep quality, and functional capacities were measured 24 hours before the intervention. The study lasted six weeks for each patient. The patients in the intervention group performed their interventions three times a week, every other day. The patients were checked by calling every week by phone. Pain, fatigue, sleep quality, and functional capacity of each patient were measured within one week at the latest, after the end of the practices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Followed up with a diagnosis of RA for at least 1 year,
* VAS pain score of 5 and above,
* Volunteer to participate in the research,
* Disease activity score is low-moderate (DAS28 < 5.1),
* Patients receiving active treatment (corticosteroid, non-steroidal anti-inflammatory, disease-modifying antirheumatic drugs) for the last 3 months were included in the study.

Exclusion Criteria:

* - Comorbidity (active malignancy, heart failure or symptomatic ischemic heart disease, severe lung disease, neurologic disease that impairs mobility, uncontrolled thyroid disease, diabetes mellitus)
* Recent injury or major surgery (within 6 months prior to enrollment)
* E-joint replacement surgery is planned,
* Acute infection, fever or vascular disease in the lower and upper extremities,
* The integrity of the skin on the hands and feet is impaired,
* Participating in a regular physical therapy or exercise program,
* pregnant,
* Diagnosed with sleep apnea
* VAS pain score below 5,
* Disease activity score ≥ 5.1,
* Patients who did not agree to participate in the study were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | It was applied just before the interventions and six weeks after interventions. Change from baseline pain scores at the end of sixth week.
  Pain is among the main reasons for rheumatoid arthritis patients to apply to the hospital and seek medical care.
Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire | It was applied just before the interventions and six weeks after the interventions. Change from baseline fatigue scores at the end of sixth week.
  Fatigue is one of the most common symptoms experienced by rheumatoid arthritis patients and this symptom affects most patients.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | It was applied just before the interventions and six weeks after interventions. Change from baseline sleep quality scores at the end of sixth week.
  An average of 50-70% of patients with rheumatoid arthritis complain of sleep disorders such as difficulty falling asleep, decreased sleep quality, restless sleep, night waking and Excessive daytime sleepiness.
Health Assessment Questionnaire | It was applied just before the interventions and six weeks after interventions. Change from baseline health assessment scores at the end of sixth week.
  The quality of life of patients with rheumatoid arthritis is adversely affected by the symptoms they experience.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgisun Kapucu, Prof., Study Chair — Hacettepe University Faculty of Nursing
Locations (1):
- S.B.Ü Gülhane Training and Education Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aktas O, Donmez AA, Kapucu S, Cinar M. The effect of warm saltwater and warm water baths on pain, fatigue, sleep quality, and functional capacity in patients with rheumatoid arthritis: a randomized controlled study✰. BMC Complement Med Ther. 2025 Aug 12;25(1):302. doi: 10.1186/s12906-025-05050-2. PMID 40790488